CLINICAL TRIAL: NCT00808132
Title: A Double-Blind, Randomized, Placebo And Active- Controlled Efficacy And Safety Study Of The Effects Of Bazedoxifene/Conjugated Estrogens Combinations On Endometrial Hyperplasia And Prevention Of Osteoporosis In Postmenopausal Women
Brief Title: Study Evaluating The Effects Of Bazedoxifene/Conjugated Estrogens On Endometrial Safety And Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3115A1-3307; B2311009
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Menopause; Osteoporosis
Keywords: Postmenopausal Women; Bazedoxifene/Conjugated Estrogens
MeSH Terms: conditions — Osteoporosis | interventions — bazedoxifene; Estrogens, Conjugated (USP); Medroxyprogesterone Acetate; Prempro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): bazedoxifene 20 mg/conjugated estrogens 0.45 mg
  Interventions: Drug: bazedoxifene 20 mg/ conjugated estrogens 0.45 mg
- 2 (Experimental): bazedoxifene 20 mg/conjugated estrogens 0.625 mg
  Interventions: Drug: bazedoxifene 20 mg/ conjugated estrogens 0.625 mg
- 3 (Experimental): bazedoxifene 20 mg
  Interventions: Drug: bazedoxifene 20 mg
- 4 (Active Comparator): Prempro
  Interventions: Drug: conjugated estrogens 0.45 mg/ medroxyprogesterone acetate 1.5 mg
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bazedoxifene 20 mg/ conjugated estrogens 0.45 mg — One capsule, bazedoxifene 20 mg/conjugated estrogens 0.45 mg (over-encapsulated), once a day for one year.
  Arms: 1
Drug: bazedoxifene 20 mg/ conjugated estrogens 0.625 mg — One capsule, bazedoxifene 20 mg/conjugated estrogens 0.625 mg (over-encapsulated), once a day for one year.
  Arms: 2
Drug: bazedoxifene 20 mg — One capsule, bazedoxifene 20 mg (over-encapsulated), once a day for one year.
  Arms: 3
Drug: conjugated estrogens 0.45 mg/ medroxyprogesterone acetate 1.5 mg — One capsule, conjugated estrogens 0.45 mg and medroxyprogesterone 1.5 mg (over-encapsulated), once a day for one year.
  Other Names: Prempro
  Arms: 4
Drug: Placebo — One capsule, placebo (over-encapsulated), once a day for one year.
  Arms: 5

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of this investigational drug for the treatment of menopausal symptoms while protecting the endometrium (uterine lining) and preventing postmenopausal osteoporosis. Subject participation will last approximately 14.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women, aged 40 to 64 seeking treatment for menopausal symptoms
* At least 12 months of spontaneous amenorrhea, OR 6 months spontaneous amenorrhea with follicle-stimulating hormone (FSH) levels > 40 mIU/mL
* Intact Uterus

Exclusion Criteria:

* Use of oral estrogen, progestin, androgen, or selective estrogen receptor modulator (SERM) containing drug products within 8 weeks before screening
* A history or active presence of clinically important medical disease: eg. cardiovascular disease (stroke, heart attack), chronic renal or liver disease, breast cancer, etc.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1886 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (153):
- United States (122):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Boynton Beach, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Crystal River, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Miami Springs, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Meridian, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Lousiville, Kentucky
  - Pfizer Investigational Site, Bangor, Maine
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Paw Paw, Michigan
  - Pfizer Investigational Site, Saginaw, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Brooklyn Center, Minnesota
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Robbinsdale, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, North Las Vegas, Nevada
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Brick, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Port Jefferson, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Kernersville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Englewood, Ohio
  - Pfizer Investigational Site, Mayfield Heights, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Erie, Pennsylvania
  - Pfizer Investigational Site, Hopwood, Pennsylvania
  - Pfizer Investigational Site, Jenkintown, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Bluffton, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Hilton Head Island, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Watertown, South Dakota
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Denton, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Pleasant Grove, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Argentina (3):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Caba, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Australia (3):
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Perth, Western Australia
- Pfizer Investigational Site, Santiago, RM, Chile
- Colombia (3):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Denmark (3):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Ballerup Municipality
  - Pfizer Investigational Site, Vejle
- Finland (2):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Oulu
- Hungary (6):
  - Pfizer Investigational Site, Békéscsaba
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Kecskemét
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Tatabánya
- Pfizer Investigational Site, D.F, Mexico, Mexico
- New Zealand (3):
  - Pfizer Investigational Site, Dunedin, NZ
  - Pfizer Investigational Site, Wellington, NZ
  - Pfizer Investigational Site, Christchurch
- Norway (2):
  - Pfizer Investigational Site, Ålesund, Norway
  - Pfizer Investigational Site, Hamar
- Poland (4):
  - Pfizer Investigational Site, Poznan, Poland
  - Pfizer Investigational Site, Wroclaw, Poland
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw

REFERENCES:
- [Derived] Pinkerton JV, Harvey JA, Lindsay R, Pan K, Chines AA, Mirkin S, Archer DF; SMART-5 Investigators. Effects of bazedoxifene/conjugated estrogens on the endometrium and bone: a randomized trial. J Clin Endocrinol Metab. 2014 Feb;99(2):E189-98. doi: 10.1210/jc.2013-1707. Epub 2014 Jan 17. PMID 24438370
- [Derived] Pinkerton JV, Harvey JA, Pan K, Thompson JR, Ryan KA, Chines AA, Mirkin S. Breast effects of bazedoxifene-conjugated estrogens: a randomized controlled trial. Obstet Gynecol. 2013 May;121(5):959-968. doi: 10.1097/AOG.0b013e31828c5974. PMID 23635731
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3115A1-3307&StudyName=Study%20Evaluating%20The%20Effects%20Of%20Bazedoxifene/Conjugated%20Estrogens%20On%20Endometrial%20Safety%20And%20Postmenopausal%20Osteoporosis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This main study also included 3 sub-studies only for the purpose of the assessment of relevant parameters: breast density sub-study, osteoporosis sub-study (OSS), and sleep sub-study. A participant could participate in more than 1 sub-study.
Groups:
- Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg: Bazedoxifene 20 milligram (mg), conjugated estrogens 0.45 mg tablets-in-capsule orally once daily at approximately the same time each day continuously for 1 year.
- Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg: Bazedoxifene 20 mg, conjugated estrogens 0.625 mg tablets-in-capsule orally once daily at approximately the same time each day continuously for 1 year.
- Bazedoxifene 20 mg: Bazedoxifene 20 mg tablet-in-capsule orally once daily at approximately the same time each day continuously for 1 year.
- Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg: Conjugated estrogens 0.45 mg, medroxyprogesterone acetate 1.5 mg tablets-in-capsule orally once daily at approximately the same time each day continuously for 1 year.
- Placebo: Placebo capsule matched to bazedoxifene/conjugated estrogen or bazedoxifene alone or conjugated estrogen/medroxyprogesterone acetate tablets-in-capsule orally once daily at approximately the same time each day continuously for 1 year.
Period: Overall Study
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Started | 455 | 481 | 239 | 228 | 483
Treated | 445 | 474 | 230 | 220 | 474
Completed | 357 | 393 | 185 | 159 | 383
Not Completed | 98 | 88 | 54 | 69 | 100
Not completed — Adverse Event | 34 | 33 | 16 | 31 | 33
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 8 | 10 | 11 | 8 | 9
Not completed — Protocol Violation | 8 | 9 | 4 | 9 | 5
Not completed — Withdrawal by Subject | 27 | 18 | 2 | 7 | 16
Not completed — Other | 6 | 4 | 6 | 2 | 15
Not completed — Randomized, but not treated | 10 | 7 | 9 | 8 | 9
Not completed — Unsatisfactory response | 5 | 6 | 6 | 4 | 12

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo | Total
Number analyzed (Participants) | 445 | 474 | 230 | 220 | 474 | 1843
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.43 (4.02) | 53.89 (4.00) | 54.07 (4.01) | 54.15 (4.50) | 54.19 (4.07) | 54.15 (4.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 445 | 474 | 230 | 220 | 474 | 1843
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endometrial Hyperplasia at Month 12: Main Study
Description: Endometrial hyperplasia was assessed by endometrial biopsies. All endometrial biopsies were read centrally by 2 primary pathologists. If both the pathologists disagreed on the presence of hyperplasia, a third pathologist was consulted. Results were summarized for two definitions of hyperplasia (simple hyperplasia with or without atypia or complex hyperplasia with or without atypia); definition 1: participants were considered to have a diagnosis of hyperplasia when the 3 pathologists disagreed but at least 1 pathologist determined hyperplasia; definition 2: participants were considered to have a diagnosis of hyperplasia if at least 2 of the 3 pathologists agreed on the diagnosis.
Time Frame: Month 12
Population: Efficacy evaluable (EE) population included all randomized participants who took at least 1 dose of study drug, who had a screening endometrial biopsy with readings by at least 2 blinded central pathologists, had a biopsy during Month 12, or had hyperplasia diagnosed before Month 12 and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 335 | 368 | 169 | 149 | 354
Percentage of Participants
  Definition 1 | 0.30 [NA to 1.41] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.54 [NA to 1.70] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.00 [NA to 1.76] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.00 [NA to 1.99] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.85 [NA to 2.18] — Only upper limit of 95% confidence interval (1-sided) was calculated.
  Definition 2 | 0.30 [NA to 1.41] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.27 [NA to 1.28] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.00 [NA to 1.76] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.00 [NA to 1.99] — Only upper limit of 95% confidence interval (1-sided) was calculated. | 0.28 [NA to 1.33] — Only upper limit of 95% confidence interval (1-sided) was calculated.

2. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Lumbar Spine at Month 12: Osteoporosis Sub-Study
Description: BMD measurements of the anteroposterior lumbar spine were acquired by using dual-energy x-ray absorptiometry (DXA) scans, twice at Month 12 for a subset of participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. Mean percentage change from baseline of the 2 readings were reported.
Time Frame: Baseline, Month 12
Population: Modified Intent-to-Treat (MITT) population included all randomized participants who met inclusion criteria for osteoporosis sub-study, who had taken at least 1 dose of the study drug, and had a baseline and at least 1 post baseline value. Last Observation Carried Forward (LOCF) method was used to impute missing values.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 119 | 139 | 56 | 59 | 139
Percent Change | 0.24 (0.29) | 0.60 (0.27) | 0.07 (0.40) | 1.30 (0.39) | -1.28 (0.28)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Analysis of covariance (ANCOVA) model was used with treatment and region as main effects and baseline BMD and years since menopause as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares (LS) Mean Difference = 1.51, 95% CI 2-sided [0.822 to 2.201]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; ANCOVA model was used with treatment and region as main effects and baseline BMD and years since menopause as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.87, 95% CI 2-sided [1.209 to 2.533]

3. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Lumbar Spine at Month 6: Osteoporosis Sub-Study
Description: BMD measurements of the anteroposterior lumbar spine were acquired by using DXA scans, twice at Month 6 for a subset of participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. Mean percentage change from baseline of the 2 readings were reported.
Time Frame: Baseline, Month 6
Population: MITT population included all randomized participants who met inclusion criteria for osteoporosis sub-study, who had taken at least 1 dose of the study drug, and had baseline and at least 1 post baseline value. LOCF method was used to impute missing values. Here "N" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 115 | 136 | 55 | 58 | 135
Percent Change | 0.12 (0.28) | 0.51 (0.26) | 0.00 (0.39) | 0.64 (0.37) | -0.68 (0.27)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.017, ANCOVA; LS Mean Difference = 0.80, 95% CI 2-sided [0.139 to 1.470]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.19, 95% CI 2-sided [0.556 to 1.830]

4. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Total Hip at Month 6, 12: Osteoporosis Sub-Study
Description: BMD measurements of the total hip were acquired by using DXA scans, twice at Month 6 and 12 for a subset of participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. Mean percentage change from baseline of the 2 readings were reported.
Time Frame: Baseline, Month 6, Month 12
Population: MITT for osteoporosis sub-study. LOCF method was used to impute missing values. Here "n" signifies participants who were evaluable at specified time points for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 119 | 139 | 56 | 59 | 139
Percent Change
  Change at Month 6 (n=117, 136, 55, 57, 134) | 0.43 (0.18) | 0.66 (0.17) | 0.32 (0.25) | 0.45 (0.24) | -0.90 (0.17)
  Change at Month 12 (n=119, 139, 56, 59, 139) | 0.50 (0.20) | 0.89 (0.18) | 0.47 (0.27) | 0.71 (0.26) | -0.72 (0.18)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Month 6: ANCOVA model was used with treatment and region as main effects and baseline BMD and years since menopause as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.32, 95% CI 2-sided [0.901 to 1.742]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Month 12: ANCOVA model was used with treatment and region as main effects and baseline BMD and years since menopause as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.21, 95% CI 2-sided [0.756 to 1.671]
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.56, 95% CI 2-sided [1.152 to 1.962]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.60, 95% CI 2-sided [1.164 to 2.044]

5. Secondary Outcome: Percentage of Participants With Cumulative Amenorrhea: Main Study
Description: Cumulative amenorrhea was defined as the absence of any bleeding or spotting for cumulative 4-week periods throughout 1-year study.
Time Frame: Day 1 up to Day 364
Population: MITT population included all randomized participants who received at least 1 dose of the study drug, and had at least 1 day of on-therapy bleeding data. Here "N" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 355 | 390 | 187 | 158 | 379
Percentage of Participants | 87.89 | 84.87 | 82.35 | 54.43 | 83.91
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Test type: Superiority or Other; p = 0.138, Fisher Exact
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Test type: Superiority or Other; p = 0.765, Fisher Exact
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 5: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

6. Secondary Outcome: Percent Change From Baseline in Breast Density at Month 12: Breast Density Sub-Study
Description: Breast density was assessed by digitalized mammograms which were centrally read by a single radiologist using specifically-developed software. Breast density was assessed for subset of participants who entered the breast density sub-study
Time Frame: Baseline, Month 12
Population: Per-Protocol (PP) population included all randomized participants who met inclusion criteria for breast density sub-study, who had a baseline and at least 1 post-baseline breast density evaluation and did not have substantial protocol violations. Here "N" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 186 | 190 | 97 | 68 | 181
Percent Change | -0.38 (0.22) | -0.45 (0.22) | -0.25 (0.30) | 1.60 (0.35) | -0.32 (0.23)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.832, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.632 to 0.509]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.651, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.696 to 0.436]

7. Secondary Outcome: Percent Change From Baseline in Bone Turnover Markers (BTMs) at Month 6 and Month 12: Osteoporosis Sub-Study
Description: Bone turnover is the removal of old bone from the body and its replacement by new bone. Bone turnover markers included serum osteocalcin, C-telopeptide, and procollagen type 1 N-propeptide (P1NP), were measured at Month 6 and Month 12 for a subset of participants who entered the osteoporosis substudy. Blood samples were collected to evaluate bone turnover markers levels.
Time Frame: Baseline, Month 6, 12
Population: MITT for osteoporosis substudy. Here "N" signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at specified time points for each arm respectively.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 115 | 136 | 57 | 56 | 134
Percent Change
  Osteocalcin: Month 6 (n=115, 136, 56, 56, 134) | -25.21 [-33.79 to -14.00] | -27.79 [-38.12 to 15.31] | -15.60 [-22.48 to -6.75] | -25.34 [-38.37 to -9.65] | -3.19 [-15.32 to 10.21]
  Osteocalcin: Month 12 (n=104, 127, 52, 50, 125) | -30.46 [-40.77 to -18.79] | -37.02 [-46.87 to -23.50] | -16.05 [-33.67 to 2.13] | -32.79 [-48.90 to -13.03] | -5.28 [-19.29 to 11.16]
  C-Telopeptide: Month 6 (n=115, 136, 56, 56, 133) | -34.16 [-48.76 to -17.35] | -41.41 [-58.94 to -25.00] | -29.37 [-40.81 to -8.23] | -54.05 [-68.67 to -34.66] | -10.17 [-26.57 to 8.62]
  C-Telopeptide: Month 12 (n=104, 127, 52,50,124) | -40.86 [-55.74 to -24.04] | -50.06 [-63.47 to -29.90] | -27.39 [-49.55 to 0.74] | -52.56 [-69.17 to -26.58] | -5.52 [-30.37 to 19.93]
  P1NP: Month 6 (n=114,135, 57, 56, 133) | -33.73 [-43.68 to -18.26] | -30.26 [-48.52 to -14.16] | -17.38 [-33.86 to -2.53] | -39.99 [-51.66 to -14.73] | 5.99 [-18.77 to 12.77]
  P1NP: Month 12 (n=103, 127, 53, 50, 125) | -42.38 [-49.71 to -24.16] | -43.58 [-58.66 to -24.91] | -23.97 [-40.42 to -7.33] | -50.19 [-62.91 to -20.83] | -11.13 [-26.66 to 6.60]
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Osteocalcin: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Bazedoxifene 20 mg; Osteocalcin: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0074, ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Osteocalcin: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Bazedoxifene 20 mg; Osteocalcin: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Osteocalcin: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Bazedoxifene 20 mg; Osteocalcin: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Osteocalcin: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Bazedoxifene 20 mg; Osteocalcin: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg vs Placebo; Osteocalcin: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg vs Placebo; Osteocalcin: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0016, ANCOVA
Statistical Analysis 11: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Osteocalcin: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 12: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Osteocalcin: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; C-Telopeptide: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Bazedoxifene 20 mg; C-Telopeptide: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.1058, ANCOVA
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; C-Telopeptide: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Bazedoxifene 20 mg; C-Telopeptide: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0024, ANCOVA
Statistical Analysis 17: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; C-Telopeptide: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 18: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Bazedoxifene 20 mg; C-Telopeptide: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; C-Telopeptide: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 20: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Bazedoxifene 20 mg; C-Telopeptide: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg vs Placebo; C-Telopeptide: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 22: Comparison: Bazedoxifene 20 mg vs Placebo; C-Telopeptide: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0012, ANCOVA
Statistical Analysis 23: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; C-Telopeptide: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 24: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; C-Telopeptide: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 25: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; P1NP: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Bazedoxifene 20 mg; P1NP: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0029, ANCOVA
Statistical Analysis 27: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; P1NP: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 28: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Bazedoxifene 20 mg; P1NP: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0046, ANCOVA
Statistical Analysis 29: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; P1NP: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 30: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Bazedoxifene 20 mg; P1NP: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0043, ANCOVA
Statistical Analysis 31: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; P1NP: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 32: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Bazedoxifene 20 mg; P1NP: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 33: Comparison: Bazedoxifene 20 mg vs Placebo; P1NP: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p = 0.0016, ANCOVA
Statistical Analysis 34: Comparison: Bazedoxifene 20 mg vs Placebo; P1NP: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 35: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; P1NP: Month 6, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 36: Comparison: Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; P1NP: Month 12, ANCOVA model was used with treatment and region as factors, and baseline as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA

8. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Scale at Baseline: Sleep Sub-Study
Description: Participant-rated questionnaire to assess sleep quality and quantity. Consists of 12-item questionnaires answered on a range of 1 to 6 for questions (Q) 3 to 12, 1 to 5 for Q1 (some questions are reversed so that a high score reflects more of the attributes); and Q2 answered on 0 to 24. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range* 100); total score range: 0 to 100; higher score = greater intensity of attribute. The items contribute to each scale and are averaged to create the 7 scale scores and a sleep quantity scale. Scales with at least one item answered was used to generate a scale score. Scales include; sleep disturbance (SD), snoring, awaken short of breath (ASoB) or with a headache (H), somnolence, sleep adequacy (SA), sleep problem index (SPI) I and II (range: 0-100) and sleep quantity (SQ [range 0 to 24]). Except for sleep quantity, higher scores=greater impairment.
Time Frame: Baseline
Population: MITT population included all randomized participants who met inclusion criteria for sleep sub-study and had baseline and at least 1 post-baseline evaluation for the respective endpoint. Here N = maximum number of participants who were evaluable for this outcome and n = participants who were evaluable at specified time points for each arm.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 112 | 121 | 47 | 52 | 111
Units on a Scale
  SD (n=112, 121, 47, 52, 111) | 48.9 (22.9) | 48.2 (21.7) | 50.5 (24.4) | 50.4 (21.1) | 47.8 (24.6)
  Snoring (n=110, 121, 47, 51, 108) | 32.1 (30.1) | 27.6 (26.9) | 37.9 (30.7) | 33.1 (29.6) | 34.4 (30.5)
  ASoB or H (n=112, 121, 47,52,111) | 12.5 (19.2) | 11.9 (19.4) | 13.2 (20.1) | 13.1 (20.2) | 12.1 (20.4)
  Somnolence (n=112, 121, 47, 52, 111) | 36.3 (21.6) | 30.0 (20.1) | 34.6 (23.5) | 28.7 (19.4) | 31.2 (19.2)
  SA (n=112, 121, 47, 52, 111) | 39.3 (24.3) | 41.7 (23.9) | 37.4 (23.2) | 36.5 (20.6) | 40.3 (23.6)
  SPI I (n=112, 121, 47, 52, 111) | 44.5 (17.3) | 42.0 (16.7) | 44.7 (18.2) | 44.9 (16.0) | 43.4 (18.1)
  SPI II (n=112, 121, 47, 52, 111) | 45.5 (17.2) | 43.2 (16.8) | 46.4 (18.0) | 45.2 (16.1) | 43.7 (18.3)
  SQ (n=111, 121, 47, 52, 111) | 6.2 (1.1) | 6.1 (1.1) | 5.9 (1.1) | 6.2 (1.3) | 6.2 (1.1)

9. Other Pre Specified Outcome: Percentage of Participants With Breast Tenderness
Description: Percentage of participants who reported at least 1 day of breast tenderness during each 4-week period for 1-year on therapy was calculated.
Time Frame: Screening, Week 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 25-28, 29-32, 33-36, 37-40, 41-44, 45-48, 49-52
Population: MITT population included all randomized participants who took 1 dose of study drug and had at least 20 days of data available at screening and at least 20 continuous days of data in at least one 4-week interval after baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 429 | 449 | 220 | 206 | 457
Percentage of Participants
  Screening (n=429, 449, 220, 206, 457) | 6.29 | 6.46 | 4.55 | 7.28 | 6.56
  Week 1-4 (n=426, 449, 220, 205, 457) | 9.39 | 9.13 | 5.91 | 20.49 | 8.32
  Week 5-8 (n=423, 447, 216, 202, 456) | 8.04 | 6.94 | 7.87 | 24.26 | 8.55
  Week 9-12 (n=412, 439, 212, 196, 447) | 5.83 | 7.97 | 6.60 | 23.98 | 5.37
  Week 13-16 (n=411, 433, 208, 193, 440) | 7.06 | 8.31 | 8.65 | 21.24 | 5.91
  Week 17-20 (n=395, 412, 197, 181, 420) | 4.05 | 4.37 | 6.09 | 17.13 | 4.29
  Week 21-24 (n=391, 410, 195, 180, 416) | 4.60 | 3.90 | 5.64 | 15.00 | 4.33
  Week 25-28 (n=389, 409, 193, 179, 416) | 3.08 | 5.62 | 4.15 | 15.64 | 4.09
  Week 29-32 (n=372, 403, 190, 171, 401) | 4.57 | 3.97 | 1.58 | 15.20 | 2.00
  Week 33-36 (n=369, 401, 188, 168, 395) | 2.98 | 3.49 | 3.19 | 12.50 | 2.28
  Week 37-40 (n=369, 399, 187, 166, 390) | 4.07 | 4.01 | 2.67 | 12.05 | 3.08
  Week 41-44 (n=359, 384, 184, 159, 382) | 3.62 | 2.60 | 1.63 | 9.43 | 2.62
  Week 45-48 (n=354, 382, 184, 157, 379) | 3.67 | 3.14 | 2.17 | 10.83 | 3.17
  Week 49-52 (n=353, 380, 183, 156, 376) | 3.12 | 2.89 | 1.64 | 9.62 | 2.66
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 1-4: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.546, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 5-8: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.821, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 9-12: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.698, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 13-16: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.446, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 17-20: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.892, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 21-24: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.810, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 25-28: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.473, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 29-32: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.030, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 33-36: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.453, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 37-40: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.391, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 41-44: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.407, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 45-48: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.644, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 49-52: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.666, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 1-4: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.641, Cochran-Mantel-Haenszel
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 5-8: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.361, Cochran-Mantel-Haenszel
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 9-12: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.100, Cochran-Mantel-Haenszel
Statistical Analysis 17: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 13-16: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.142, Cochran-Mantel-Haenszel
Statistical Analysis 18: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 17-20: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.906, Cochran-Mantel-Haenszel
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 21-24: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.798, Cochran-Mantel-Haenszel
Statistical Analysis 20: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 25-28: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.258, Cochran-Mantel-Haenszel
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 29-32: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.058, Cochran-Mantel-Haenszel
Statistical Analysis 22: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 33-36: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.230, Cochran-Mantel-Haenszel
Statistical Analysis 23: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 37-40: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.360, Cochran-Mantel-Haenszel
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 41-44: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.892, Cochran-Mantel-Haenszel
Statistical Analysis 25: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 45-48: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.912, Cochran-Mantel-Haenszel
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 49-52: Cochran-Mantel-Haenszel test was stratified by baseline value; Test type: Superiority or Other; p = 0.791, Cochran-Mantel-Haenszel

10. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale at Month 3: Sleep Sub-Study
Description: as for outcome 8
Time Frame: Baseline, Month 3
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 112 | 121 | 47 | 52 | 111
Units on a Scale
  SD (n=112, 121, 47, 52, 111) | -17.27 (2.01) | -18.18 (1.94) | -11.64 (2.94) | -18.01 (2.79) | -14.34 (2.01)
  Snoring (n=110, 121, 47, 51, 108) | -5.86 (1.83) | -5.38 (1.76) | -2.54 (2.67) | -2.90 (2.55) | -2.71 (1.84)
  ASoB or H (n=112,121,47,52,111) | -4.26 (1.41) | -5.81 (1.35) | -3.12 (2.06) | -3.62 (1.95) | -3.63 (1.40)
  Somnolence (n=112,121,47,52,111) | -10.54 (1.53) | -9.72 (1.48) | -6.12 (2.25) | -7.36 (2.14) | -10.55 (1.53)
  SA (n=112, 121, 47, 52, 111) | 14.22 (2.40) | 14.30 (2.32) | 9.10 (3.52) | 15.10 (3.34) | 11.46 (2.40)
  SPI I (n=112, 121, 47, 52, 111) | -13.19 (1.51) | -13.99 (1.46) | -8.92 (2.21) | -13.71 (2.09) | -11.84 (1.50)
  SPI II (n=112, 121, 47, 52,111) | -14.01 (1.51) | -14.53 (1.46) | -9.64 (2.21) | -14.12 (2.10) | -12.04 (1.51)
  SQ (n=111, 121, 47, 52, 111) | 0.28 (0.10) | 0.44 (0.09) | 0.32 (0.14) | 0.41 (0.13) | 0.36 (0.10)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Sleep disturbance: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.253, ANCOVA; LS Mean Difference = -2.93, 95% CI 2-sided [-7.96 to 2.10]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Sleep disturbance: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.127, ANCOVA; LS Mean Difference = -3.84, 95% CI 2-sided [-8.78 to 1.10]
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Snoring: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.180, ANCOVA; LS Mean Difference = -3.15, 95% CI 2-sided [-7.76 to 1.46]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Snoring: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.247, ANOVA; LS Mean Difference = -2.67, 95% CI 2-sided [-7.19 to 1.85]
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; ASoB: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.726, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-4.15 to 2.90]
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; ASoB: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.218, ANCOVA; LS Mean Difference = -2.17, 95% CI 2-sided [-5.63 to 1.29]
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Somnolence: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.996, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-3.85 to 3.87]
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Somnolence: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.665, ANCOVA; LS Mean DIfference = 0.83, 95% CI 2-sided [-2.94 to 4.60]
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Sleep adequacy: Month 3, ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.368, ANOVA; LS Mean Difference = 2.76, 95% CI 2-sided [-3.26 to 8.78]
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Sleep adequacy: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.345, ANCOVA; LS Mean Difference = 2.84, 95% CI 2-sided [-3.07 to 8.75]
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Sleep problem index I: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.482, ANCOVA; LS Mean Difference = -1.35, 95% CI 2-sided [-5.12 to 2.42]
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Sleep problem index I: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.254, ANCOVA; LS Mean DIfference = -2.15, 95% CI 2-sided [-5.86 to 1.55]
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Sleep problem index II: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.308, ANCOVA; LS Mean Difference = -1.97, 95% CI 2-sided [-5.76 to 1.82]
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Sleep problem index II: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.190, ANCOVA; LS Mean Difference = -2.48, 95% CI 2-sided [-6.20 to 1.23]
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Sleep quantity: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.550, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.32 to 0.17]
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Sleep quantity: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.477, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.15 to 0.32]

11. Secondary Outcome: Menopause-Specific Quality of Life (MENQOL) Score at Baseline: Sleep Sub-Study
Description: MENQOL questionnaire assessed how bothered participants were due to menopause. It consists of 29 items divided into 4 domains: vasomotor function (3 items), psychosocial function (7 items), physical function (16 items), and sexual function (3 items). Each item scores a range from 1 to 8, with 1 indicating that the participant did not experience the symptom or problem, 8 indicating that the participant was extremely bothered by the symptom or problem. The total score for each domain is the average of item scores and ranged from 1 to 8 with higher score indicating worsening of symptoms. The MENQOL total score is the mean of these 4 domain scores and ranged from 1 to 8 with higher score indicating worsening of symptoms.
Time Frame: Baseline
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 111 | 121 | 47 | 52 | 112
Units on a Scale
  Vasomotor function (n=111, 121, 47, 52, 112) | 5.40 (1.564) | 5.60 (1.468) | 5.87 (1.246) | 5.65 (1.620) | 5.62 (1.596)
  Psychosocial function (n=111, 121, 47, 52, 112) | 3.46 (1.716) | 3.41 (1.628) | 3.49 (1.663) | 3.48 (1.793) | 3.22 (1.522)
  Physical function (n=111, 121, 47, 52, 112) | 3.74 (1.377) | 3.58 (1.385) | 3.96 (1.475) | 3.74 (1.409) | 3.58 (1.445)
  Sexual function (n=110, 121, 47, 52, 112) | 3.74 (2.200) | 3.63 (2.182) | 4.05 (2.265) | 3.73 (2.238) | 3.83 (2.243)
  MENQOL Total Score (n=110, 121, 47, 52, 112) | 4.07 (1.227) | 4.05 (1.246) | 4.34 (1.156) | 4.15 (1.314) | 4.06 (1.155)

12. Secondary Outcome: Change From Baseline in Menopause-Specific Quality of Life (MENQOL) Score at Month 3: Sleep Sub-Study
Description: as for outcome 11
Time Frame: Baseline, Month 3
Population: MITT population included all randomized participants who met inclusion criteria for sleep sub-study and had baseline and at least 1 post-baseline evaluation for the respective endpoint. Here "N": maximum number of participants who were evaluable for this outcome and "n": participants who were evaluable at specified time points for each arm.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 111 | 121 | 47 | 52 | 112
Units on a Scale
  Vasomotor function (n=111, 121, 47, 52, 112) | -2.37 (0.17) | -2.75 (0.17) | -1.25 (0.25) | -3.19 (0.24) | -1.45 (0.17)
  Psychosocial function (n=111, 121, 47, 52, 112) | -0.67 (0.12) | -0.84 (0.12) | -0.47 (0.18) | -0.83 (0.17) | -0.74 (0.12)
  Physical function (n=111, 121, 47, 52, 112) | -0.92 (0.10) | -1.11 (0.10) | -0.67 (0.15) | -0.76 (0.14) | -0.87 (0.10)
  Sexual function (n=110, 121, 47, 52, 112) | -1.20 (0.16) | -1.40 (0.15) | -0.09 (0.23) | -0.76 (0.22) | -1.04 (0.16)
  MENQOL Total Score (n=110, 121, 47, 52, 112) | -1.27 (0.10) | -1.53 (0.10) | -0.63 (0.15) | -1.39 (0.14) | -1.03 (0.10)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Vasomotor function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Vasomotor function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Psychosocial function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.680, ANCOVA
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Psychosocial function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.493, ANCOVA
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Physical function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.698, ANCOVA
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Physical function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.055, ANCOVA
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Sexual function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.428, ANCOVA
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Sexual function: ANCOVA model was used with treatment and region as factors and baseline as a covariate; Test type: Superiority or Other; p = 0.071, ANCOVA

13. Secondary Outcome: Percentage of Participants With Uterine Bleeding
Description: Percentage of participants with uterine bleeding were calculated for each 4-week period for 1-year on therapy.
Time Frame: Week 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 25-28, 29-32, 33-36, 37-40, 41-44, 45-48, 49-52
Population: MITT population included all randomized participants who took at least 1 dose of the study drug, and had at least 1 day of on-therapy bleeding data. Here "N" signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at specified time points for each arm respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 440 | 468 | 229 | 216 | 470
Percentage of Participants
  Week 1-4 (n=440, 468, 229, 216, 470) | 3.86 | 6.20 | 5.68 | 20.83 | 4.68
  Week 5-8 (n=428, 458, 221, 205, 462) | 4.44 | 5.02 | 3.62 | 24.39 | 4.11
  Week 9-12 (n=417, 451, 217, 199, 452) | 2.16 | 3.55 | 2.76 | 25.63 | 4.42
  Week 13-16 (n=415, 446, 213, 196, 446) | 2.41 | 2.91 | 3.29 | 24.49 | 3.36
  Week 17-20 (n=399,426,201,184,427) | 2.26 | 2.58 | 2.49 | 18.48 | 3.51
  Week 21-24 (n=395, 424, 199, 183, 423) | 2.78 | 2.12 | 2.01 | 18.58 | 3.31
  Week 25-28 (n=393, 422, 197, 182, 420) | 2.04 | 2.13 | 1.02 | 14.84 | 3.33
  Week 29-32 (n=376, 416, 194, 173, 405) | 1.60 | 1.68 | 1.55 | 12.14 | 1.73
  Week 33-36 (n=373, 413, 192, 170, 399) | 0.54 | 2.91 | 2.08 | 12.94 | 2.26
  Week 37-40 (n=373, 411, 191, 168, 394) | 1.61 | 2.92 | 1.57 | 14.29 | 4.82
  Week 41-44 (n=363, 396, 188, 162, 386) | 1.38 | 1.26 | 0.00 | 13.58 | 1.55
  Week 45-48 (n=358, 394, 188, 160, 383) | 0.84 | 2.28 | 0.53 | 14.38 | 2.09
  Week 49-52 (n=357, 392, 187, 159, 380) | 1.68 | 1.28 | 1.07 | 8.81 | 1.58
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.624, Fisher Exact
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.868, Fisher Exact
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.087, Fisher Exact
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.425, Fisher Exact
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.307, Fisher Exact
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.689, Fisher Exact
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.285, Fisher Exact
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.065, Fisher Exact
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.014, Fisher Exact
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.226, Fisher Exact
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Placebo; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 17: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 18: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 20: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 22: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 23: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 25: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 27: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.317, Fisher Exact
Statistical Analysis 28: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.531, Fisher Exact
Statistical Analysis 29: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.610, Fisher Exact
Statistical Analysis 30: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.848, Fisher Exact
Statistical Analysis 31: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.551, Fisher Exact
Statistical Analysis 32: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.300, Fisher Exact
Statistical Analysis 33: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.299, Fisher Exact
Statistical Analysis 34: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 35: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.660, Fisher Exact
Statistical Analysis 36: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.199, Fisher Exact
Statistical Analysis 37: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.770, Fisher Exact
Statistical Analysis 38: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 39: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Placebo; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.769, Fisher Exact
Statistical Analysis 40: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 41: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 42: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 43: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 44: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 45: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 46: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 47: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 48: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 49: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 50: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 51: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 52: Comparison: Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg vs Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg | Bazedoxifene 20 mg | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Serious Adverse Events (participants affected / at risk) | 16/445 | 17/474 | 5/230 | 13/220 | 18/474
Other Adverse Events (participants affected / at risk) | 407/445 | 426/474 | 207/230 | 197/220 | 423/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg (N=445) | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg (N=474) | Bazedoxifene 20 mg (N=230) | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg (N=220) | Placebo (N=474)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 3 | 2
Benign fallopian tube neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bazedoxifene 20 mg / Conjugated Estrogens 0.45 mg (N=445) | Bazedoxifene 20 mg / Conjugated Estrogens 0.625 mg (N=474) | Bazedoxifene 20 mg (N=230) | Conjugated Estrogens 0.45mg/Medroxyprogesterone Acetate 1.5mg (N=220) | Placebo (N=474)
Abdominal discomfort (Gastrointestinal disorders) | 11 | 13 | 8 | 6 | 10
Abdominal distension (Gastrointestinal disorders) | 9 | 13 | 4 | 7 | 13
Abdominal pain (Gastrointestinal disorders) | 23 | 34 | 15 | 13 | 31
Abdominal pain lower (Gastrointestinal disorders) | 5 | 5 | 6 | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 21 | 21 | 7 | 9 | 17
Constipation (Gastrointestinal disorders) | 20 | 25 | 14 | 14 | 20
Diarrhoea (Gastrointestinal disorders) | 33 | 36 | 13 | 13 | 24
Dyspepsia (Gastrointestinal disorders) | 24 | 13 | 9 | 11 | 14
Flatulence (Gastrointestinal disorders) | 13 | 9 | 2 | 4 | 11
Gastritis (Gastrointestinal disorders) | 4 | 2 | 5 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4 | 1 | 0 | 12
Nausea (Gastrointestinal disorders) | 32 | 29 | 8 | 11 | 26
Toothache (Gastrointestinal disorders) | 21 | 20 | 8 | 8 | 17
Vomiting (Gastrointestinal disorders) | 14 | 10 | 7 | 6 | 12
Fatigue (General disorders) | 12 | 12 | 7 | 4 | 12
Oedema peripheral (General disorders) | 10 | 4 | 3 | 4 | 5
Pain (General disorders) | 20 | 24 | 16 | 7 | 22
Pyrexia (General disorders) | 10 | 10 | 5 | 5 | 6
Seasonal allergy (Immune system disorders) | 14 | 14 | 4 | 6 | 9
Bronchitis (Infections and infestations) | 8 | 14 | 8 | 9 | 14
Cystitis (Infections and infestations) | 10 | 11 | 8 | 6 | 6
Ear infection (Infections and infestations) | 3 | 6 | 1 | 6 | 4
Gastroenteritis (Infections and infestations) | 3 | 5 | 4 | 5 | 7
Influenza (Infections and infestations) | 27 | 30 | 18 | 13 | 23
Nasopharyngitis (Infections and infestations) | 91 | 72 | 44 | 32 | 65
Sinusitis (Infections and infestations) | 42 | 37 | 19 | 12 | 33
Tooth infection (Infections and infestations) | 8 | 11 | 6 | 3 | 11
Upper respiratory tract infection (Infections and infestations) | 36 | 38 | 9 | 13 | 30
Urinary tract infection (Infections and infestations) | 30 | 20 | 14 | 5 | 33
Contusion (Injury, poisoning and procedural complications) | 7 | 3 | 4 | 4 | 15
Muscle strain (Injury, poisoning and procedural complications) | 7 | 9 | 8 | 5 | 16
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 9 | 8 | 4 | 5 | 13
Procedural pain (Injury, poisoning and procedural complications) | 26 | 36 | 6 | 14 | 30
Blood cholesterol increased (Investigations) | 10 | 5 | 7 | 1 | 7
Gamma-glutamyltransferase increased (Investigations) | 10 | 3 | 2 | 2 | 3
Low density lipoprotein increased (Investigations) | 4 | 3 | 5 | 1 | 4
Weight increased (Investigations) | 11 | 13 | 5 | 9 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 49 | 22 | 19 | 47
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 52 | 64 | 29 | 25 | 65
Muscle spasms (Musculoskeletal and connective tissue disorders) | 48 | 45 | 26 | 14 | 33
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 31 | 34 | 10 | 9 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 28 | 21 | 13 | 25
Neck pain (Musculoskeletal and connective tissue disorders) | 21 | 23 | 9 | 6 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 46 | 17 | 31 | 45
Dizziness (Nervous system disorders) | 17 | 16 | 7 | 9 | 11
Headache (Nervous system disorders) | 96 | 109 | 48 | 54 | 122
Migraine (Nervous system disorders) | 7 | 8 | 5 | 3 | 12
Sinus headache (Nervous system disorders) | 12 | 14 | 7 | 7 | 15
Anxiety (Psychiatric disorders) | 9 | 16 | 4 | 7 | 9
Depression (Psychiatric disorders) | 13 | 9 | 6 | 5 | 9
Insomnia (Psychiatric disorders) | 27 | 25 | 15 | 12 | 32
Haematuria (Renal and urinary disorders) | 6 | 5 | 7 | 1 | 8
Breast pain (Reproductive system and breast disorders) | 4 | 11 | 2 | 4 | 2
Breast tenderness (Reproductive system and breast disorders) | 17 | 19 | 5 | 26 | 18
Metrorrhagia (Reproductive system and breast disorders) | 5 | 5 | 2 | 8 | 6
Pelvic pain (Reproductive system and breast disorders) | 6 | 8 | 1 | 6 | 8
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 5 | 1 | 7 | 5
Uterine spasm (Reproductive system and breast disorders) | 11 | 6 | 6 | 7 | 8
Vaginal discharge (Reproductive system and breast disorders) | 6 | 7 | 2 | 4 | 11
Vaginal haemorrhage (Reproductive system and breast disorders) | 30 | 29 | 14 | 37 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 30 | 10 | 11 | 30
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 8 | 9 | 6 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 26 | 12 | 22 | 16
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 21 | 4 | 7 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 9 | 3 | 4 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 12 | 4 | 6 | 12
Rash (Skin and subcutaneous tissue disorders) | 8 | 15 | 4 | 6 | 5
Hot flush (Vascular disorders) | 27 | 37 | 20 | 11 | 40
Hypertension (Vascular disorders) | 15 | 9 | 4 | 6 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.